CLINICAL TRIAL: NCT07111130
Title: Prospective Interventional Study Evaluating the Modulation of Bile Acid Profiles, Gut Microbiome and Liver Health Through Lifestyle Adjustments in Individuals at High Risk of Developing Liver Cancer.
Brief Title: Restoring Bile Acid Homeostasis Via Lifestyle Adjustments to Prevent the Development of Liver Cancer
Acronym: RE-BALANCE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Perspectum (Industry); BUZUD Pte Ltd (Unknown); Asian Microbiome Library (AMiLi) Pte Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AHCC14
Record Dates: First submitted 2025-07-15; First posted 2025-08-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Liver Diseases
Keywords: Hepatocellular Carcinoma (HCC); Non-viral HCC; Interventional Study; Lifestyle Adjustments; Bile Acid, Microbiome and Liver Health Modulation
MeSH Terms: conditions — Liver Diseases; Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Patients eligible for the RE-BALANCE study will be selected from the ELEGANCE cohort based on predefined high-risk criteria, specifically a low 12-non-hydroxy/12-hydroxy bile acid ratio indicative of elevated hepatocarcinogenic risk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12-week Intervention (Experimental): 12-week lifestyle intervention.
  Interventions: Other: 12-week Lifestyle Intervention

INTERVENTIONS:
Other: 12-week Lifestyle Intervention — Eligible participants within the existing ELEGANCE cohort will undergo a structured 12-week lifestyle intervention comprising a low-carbohydrate, high-fibre dietary plan and a prescribed physical activity program targeting at least 150 minutes of moderate-intensity exercise per week. Standardized meal provision and wearable fitness tracking devices will be used to support adherence throughout the intervention period.

SUMMARY:
This is a prospective, single-arm, non-randomized interventional study nested within the existing ELEGANCE cohort. Patients eligible for the RE-BALANCE study will be selected from the ELEGANCE cohort based on predefined high-risk criteria, specifically a low 12-non-hydroxy/12-hydroxy bile acid ratio indicative of elevated hepatocarcinogenic risk.

The study comprises Baseline Assessments (Visit 1), Intervention Visits (Visit 2-8), and Follow-up Assessments (Visit 9-11).

DETAILED DESCRIPTION:
Participants will undergo a structured 12-week lifestyle intervention comprising a low-carbohydrate, high-fibre dietary plan and a prescribed physical activity program targeting at least 150 minutes of moderate-intensity exercise per week. Standardized meal provision and wearable fitness tracking devices will be used to support adherence throughout the intervention period.

Biological assessments will be conducted at baseline (Visit 1), mid-intervention (Visit 6), and end-of-intervention (Visit 9), including blood sampling for bile acid profiling and stool sampling for gut microbiome sequencing. Liver health evaluation will be conducted at baseline (Visit 1) and end-of-intervention (Visit 9) to assess patient's change in liver health. Extended biological assessments (Visit 10-11) and liver health evaluation through LMS-CT1 imaging (Visit 11) will be performed post-intervention to evaluate the sustainability of the observed changes.

Participants will continue to receive standard-of-care surveillance in parallel during the study. In the event of clinical suspicion for hepatocellular carcinoma during surveillance imaging, participants will undergo confirmatory diagnostic imaging and, if diagnosed, will be referred for standard clinical management. Participants diagnosed with HCC during the study will be withdrawn from the active intervention phase. Their data up to the point of diagnosis will be included in analysis, and they will revert to standard-of-care HCC management. Ongoing follow-up for clinical outcomes may continue under the parent ELEGANCE study framework.

The study will enrol approximately 90 high-risk NBNC patients identified from the ELEGANCE cohort. Accrual is expected to be completed within 6 to 9 months. The active intervention will last 12 weeks, with subsequent observational follow-up extending up to 12 months post-intervention to assess the durability of metabolic, microbiome, and imaging changes and monitor the incidence of hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

The following criteria are to be checked at the time of enrolment. The patient may only be included in the study if ALL of the following statements are FULFILLED:

1. The patient is an existing participant of the ELEGANCE study and shows no evidence of hepatocellular carcinoma (HCC) at the time of enrolment into RE-BALANCE.
2. Male and female patients aged 50 to 90 years at the time of informed consent are eligible. However, patients with cirrhosis may be included if they are aged 40 to 90 years.
3. Negative for hepatitis B surface antigen (HBsAg) and hepatitis C antibody
4. High-risk bile acid profile, defined as a 12-non-hydroxy/12-hydroxy bile acid ratio below the threshold determined from ELEGANCE cohort data.
5. Patient is able to comply with scheduled visits, assessments and other study procedures.
6. Patient is willing to provide informed consent before enrolment in the study.

Exclusion Criteria:

The following criteria should be checked at the time of enrolment. If ANY applies, the patient must not be included in the study:

1. Patient with confirmed diagnosis of HCC by the American Association for the Study of the Liver Disease (AASLD) imaging criteria or histology / cytology within the last 5 years.
2. Patient with Child Pugh C or decompensated cirrhosis at time of enrolment (based on the judgement of the Investigator).
3. Patient with active hepatic encephalopathy at time of enrolment.
4. Patient is known to be positive for the Human Immunodeficiency Virus (HIV).
5. Patient has chronic liver diseases apart from steatosis or compensated cirrhosis (e.g., autoimmune hepatitis, primary biliary cholangitis. etc.).
6. Uncontrolled diabetes mellitus requiring special dietary management or persistent unacceptable HbA1c levels.
7. Use of weight-loss medications (e.g., GLP-1 agonists, Orlistat) within three months prior to enrolment or planned use during the study period.
8. History of bariatric surgery or planned bariatric surgery during the study period.
9. Patient has significant comorbidities expected to limit life expectancy to less than one year, or that would render diet or exercise unsafe

   1. Diseases involving muscles, bones or joints that may impact the subjects' performance during exercise testing and exercise rehabilitation
   2. Co-morbidities that may adversely affect exercise performance
   3. Requiring an assistive aid with walking
   4. Conditions that require strict dietary restrictions or impair ability to follow dietary interventions
10. Patient has significant gastrointestinal diseases affecting nutrient absorption or requiring a special diet incompatible with study diet.
11. Pregnancy or breastfeeding
12. Current use of medications or supplements that significantly alter bile acid gastrointestinal absorption (e.g., bile acid sequestrants) that cannot be safely discontinued.
13. Patient has severe food allergies or intolerances incompatible with the provided study diet.
14. Patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the study procedures.
15. Patient is unable to provide informed consent or refuse blood taking and other investigations including LMS scans.
16. Patient has any other condition which, in the opinion of the Investigators, would make the patient unsuitable for enrolment or could interfere with completion of the study.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Hepatocarcinogenic risk change in relation to metabolomics profile. | Pre-intervention (Baseline), Post-intervention (3-month)
  Change in the bile acid profile pre- and post-intervention.
Hepatocarcinogenic risk change in relation to metagenomics profile. | Pre-intervention (Baseline), Post-intervention (3-month)
  Change in the gut microbiome alpha and beta diversity pre- and post-intervention.
Hepatocarcinogenic risk change in relation to liver health profile. | Pre-intervention (Baseline), Post-intervention (3-month)
  Change in the hepatic steatosis and fibrosis as measured by LMS-CT1 MRI pre- and post-intervention.
Sustained change in hepatocarcinogenic risk in relation to metabolomics profile. | Up to 12 months.
  Sustained change in the bile acid profile post-intervention.
Sustained change in hepatocarcinogenic risk in relation to metagenomics profile. | Up to 12 months.
  Sustained change in the gut microbiome alpha and beta diversity post-intervention.
Sustained change in hepatocarcinogenic risk in relation to liver health profile. | Up to 12 months.
  Sustained change in the hepatic steatosis and fibrosis as measured by LMS-CT1 MRI post-intervention.
Long-term HCC incidence against a matched control within the ELEGANCE cohort. | Up to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Pierce Chow, MD, PhD, Study Chair — National Cancer Centre, Singapore
Locations (14):
- Singapore (14):
  - National University Hospital, Singapore
  - SingHealth Polyclinics - Bukit Merah, Singapore
  - National Cancer Center Singapore, Singapore
  - SingHealth Polyclinics - Outram, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - SingHealth Polyclinics - Marine Parade, Singapore
  - SingHealth Polyclinics - Bedok, Singapore
  - SingHealth Polyclinics - Pasir Ris, Singapore
  - SingHealth Polyclinics - Tampines, Singapore
  - Changi General Hospital, Singapore
  - Sengkang General Hospital, Singapore
  - SingHealth Polyclinics - Sengkang, Singapore
  - SingHealth Polyclinics - Punggol, Singapore

IPD SHARING:
Plan to Share IPD: No